CLINICAL TRIAL: NCT05102331
Title: Lavender Oil Aromatherapy for The Treatment of Acute Anxiety During Bone Marrow Biopsy Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4Z21
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender Oil Aromatherapy Treatment Arm (LOA) (Experimental): Participants will complete baseline assessments including 20 minutes of questionnaires and vitals assessment, including EEG activity (baseline measured with Bispectral Index (BIS) device). Participants will be given a dental bib with three lavender oil drops and instructed to relax for 20 minutes. BP and a brief self-report measure will be obtained. BIS recordings will be collected continuously during study and biopsy.
  At procedure, participants will continue to wear bib with drops. BIS machine will stay attached and recording. Participants will be asked to verbally report pain and anxiety on visual analogue scale between the bone marrow aspirate and biopsy. EEG and heart rate (HR) will be collected continuously. An event marker and notation will indicate times when participant does something that may influence EEG activity (e.g. speak, move, etc.) or diagnostic images are taken. At procedure end, BIS device will be removed, final questionnaires administered, and vitals measured.
  Interventions: Other: Lavender Oil Aromatherapy; Procedure: BMAB procedure
- Placebo Aromatherapy Control Arm (PA) (Placebo Comparator): Participants assigned to PA Clinic staff will have the same procedures as listed in LOA arm except the oil used will be a refined jojoba oil which has no color or smell. The BMAB procedure will follow the SOC provided by the clinic. This includes warning participants of upcoming stimuli, encouraging patients to remain calm, and generally expressing empathy to participants. Participants in this group will receive the same collection of questionnaires before, during, and after the procedure as the LOA group. BP, HR, and EEG measurements will similarly be collected continuously before, during, and after the procedure.
  Interventions: Other: Placebo oil; Procedure: BMAB procedure

INTERVENTIONS:
Other: Lavender Oil Aromatherapy — Participants will be given a dental bib to wear. Three drops of the lavender oil will be placed on the fabric of the bib and the participant will be instructed to relax for 20 minutes.
  The lavender oil is produced by doTERRA and has Gas Chromatography Mass Spectrometry analysis showing 35.66% linalool without any contaminants
  Arms: Lavender Oil Aromatherapy Treatment Arm (LOA)
Other: Placebo oil — Participants will be given a dental bib to wear. Three drops of the placebo oil will be placed on the fabric of the bib and the participant will be instructed to relax for 20 minutes.
  Refined jojoba oil which has no color or smell
  Arms: Placebo Aromatherapy Control Arm (PA)
Procedure: BMAB procedure — SOC BMAB procedure. The procedure takes approximately 20 minutes to complete and is performed on the posterior superior iliac crest of the pelvic bone. Between 5 and 10 mL of 1% lidocaine will be injected into the site of the BMAB 5 minutes prior to the procedure beginning. No systemic premedications will be allowed including opioids or benzodiazepines. If during the procedure, participants continue to report severe anxiety or pain, the practitioner may consider providing 1mg of lorazepam or morphine as a rescue medication. The aspirate needle and core biopsy needle will be the standard needle provided by the BMAB kit

SUMMARY:
The purpose of this study is to assess the effectiveness of lavender oil as compared to standard of care (SOC) to relieve anxiety in participants undergoing a bone marrow aspirate and biopsy procedure

DETAILED DESCRIPTION:
Bone marrow aspiration and biopsy (BMAB) is a primarily outpatient procedure that is used to aid the diagnosis of hematological diseases. During the BMAB, local anesthesia is used however, many recipients still commonly report pain. Poorly-controlled pain has been shown to have adverse, long-lasting psychological effects and those receiving BMAB are generally significantly anxious and concerned about pain when undergoing this procedure. Previous clinical studies suggest that lavender oil aromatherapy is effective in lowering anxiety experienced by participants. It will be hypothesized that lavender oil aromatherapy will demonstrate benefit to participants suffering from anxiety during the BMAB procedure.

Participants who are undergoing BMAB and meet the inclusion criteria will be randomized to either receive aromatherapy via lavender oil before and during the duration of the BMAB, or to a SOC arm.

The primary objective of this study is to assess the efficacy of lavender oil aromatherapy as compared to placebo aromatherapy to relieve acute anxiety in participants undergoing a BMAB procedure

Secondary objectives of this study are:

To assess the efficacy of lavender oil aromatherapy as compared to placebo aromatherapy to relieve acute anxiety in participants undergoing a BMAB procedure

To determine the feasibility of utilizing lavender oil aromatherapy during BMAB in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and sign a written informed consent document, and be willing to follow protocol requirements
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Willingness to comply with all study interventions of lavender oil aromatherapy
* Anxiety >3 on a 0-10 visual analog scale regarding the bone marrow biopsy/aspirate procedure

Exclusion Criteria:

* Allergy to lavender oil
* Mental incapacitation (ex. stroke, brain metastasis etc.) that would cause inability to follow directions, in the opinion of the investigators
* Ongoing uncontrolled active psychiatric condition that would interfere in the conduct of the study (e.g., mood disorders, anxiety, psychosis disorders, or substance use), as determined by the patient's primary cancer team.
* If a patient has a history of a psychiatric disorder, we will contact their primary cancer team to determine if their condition is controlled or uncontrolled, and if it will interfere with the study.
* Currently pregnant
* Recent changes in the past 2 weeks to medications prescribed for pain or anxiety

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Anxiety scores from post-procedure questionnaire | Within fifteen minutes post-BMAB
  Efficacy of LOA as compared to SOC to relieve acute anxiety in participants undergoing a BMAB procedure will be assessed by comparing anxiety scores from a post-procedure questionnaire that asks "What was the highest level of anxiety that you experienced during the procedure?"
  The primary analysis will compare difference scores from this anxiety score between the two groups using the Wilcoxon-Mann-Whitney test (Higher the score more is the anxiety).
State-Trait Anxiety Inventory (STAI) scores - Baseline | Within fifteen minutes pre-BMAB
  The STAI measure one's conscious awareness at two extremes of anxiety affect, labeled state anxiety (A-state), and trait anxiety (A-trait), respectively.
  The STAI includes 20 questions about how the participant is feeling (e.g. I feel worried), each ranging from 1 to 4, with 1 indicating "not at all" and 4 indicating "very much so". Full scale ranges from 40 to 160, with higher STAI scores suggesting higher levels of anxiety.
  This study will use STAI at baseline and then the state anxiety inventory short form (SAI-SF) for the subsequent time points.
SAI-SF scores | Within fifteen minutes post-BMAB
  The SAI-SF utilizes six questions from the STAI state questionnaire to assess state anxiety and has shown similar results to the full form. Scores range from 6 to 24, with higher scores indicating worse anxiety.
  Questions relate to feeling: calm, tense, upset, relaxed, content and worried

SECONDARY OUTCOMES:
Pain scores based on the Brief Pain Inventory Short Form (BPI-SF) | Within fifteen minutes pre-BMAB
  Efficacy of LOA to relieve acute pain as measured by BPI-SF scores.
  Item 1: Yes/No question assessing if participants are currently experiencing pain other than minor headache, sprain, or toothache.
  Item 2: Aks participants to indicate on a whole body diagram the exact location of pain.
  Items 3-6: Measure severity of pain on a 0-10 numeric scale, with 0 indicating no pain and 10 indicating pain as bad as you can imagine Item 7: Asks "what treatment or medications are you receiving for your pain?" Item 8: Assesses relief from pain treatments or medications within the last 24 hours, scored by "percent of relief received" from 0% to 100%, at 10% increments, with 0% indicating no relief, and 100% indicating complete relief Item 9 includes 7 sub-ratings regarding the impact that pain within the previous 24 hours on quality of life. Each sub-rating is scored from 0 to 10 with 0 indicating that pain does not interfere, and 10 indicating pain completely interferes.
Pain scores based on the BPI-SF | Within fifteen minutes post-BMAB
  Efficacy of LOA to relieve acute pain as measured by BPI-SF scores.
  Item 1: Yes/No question assessing if participants are currently experiencing pain other than minor headache, sprain, or toothache.
  Item 2: Aks participants to indicate on a whole body diagram the exact location of pain.
  Items 3-6: Measure severity of pain on a 0-10 numeric scale, with 0 indicating no pain and 10 indicating pain as bad as you can imagine Item 7: Asks "what treatment or medications are you receiving for your pain?" Item 8: Assesses relief from pain treatments or medications within the last 24 hours, scored by "percent of relief received" from 0% to 100%, at 10% increments, with 0% indicating no relief, and 100% indicating complete relief Item 9 includes 7 sub-ratings regarding the impact that pain within the previous 24 hours on quality of life. Each sub-rating is scored from 0 to 10 with 0 indicating that pain does not interfere, and 10 indicating pain completely interferes.
Pain scores based on Edmonton Symptom Assessment Score (ESAS) | Within fifteen minutes pre-BMAB
  Average pain symptom scores as measured by ESAS
  The ESAS measures responses to 10 common symptoms (pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, feelings of well-being, and other symptom). Participants rate the intensity of symptoms during the last 24 hours on 0 to 10 numerical scales from 0 no symptom to 10 worst possible symptoms.
Pain scores based on ESAS | Within fifteen minutes post-BMAB
  Average pain symptom scores as measured by ESAS
  The ESAS measures responses to 10 common symptoms (pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, feelings of well-being, and other symptom). Participants rate the intensity of symptoms during the last 24 hours on 0 to 10 numerical scales from 0 no symptom to 10 worst possible symptoms.
Anxiety scores based on ESAS | Within fifteen minutes pre-BMAB
  Average anxiety symptom scores as measured by ESAS
  The ESAS measures responses to 10 common symptoms (pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, feelings of well-being, and other symptom). Participants rate the intensity of symptoms during the last 24 hours on 0 to 10 numerical scales from 0 no symptom to 10 worst possible symptoms.
  A mixed effect regression model with the anxiety scores from the ESAS will be fit to assess association between groups and outcomes. The study team will also test for time effects and for a group by time interaction effect.
Anxiety scores based on ESAS | Within fifteen minutes post-BMAB
  Average anxiety symptom scores as measured by ESAS
  The ESAS measures responses to 10 common symptoms (pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, feelings of well-being, and other symptom). Participants rate the intensity of symptoms during the last 24 hours on 0 to 10 numerical scales from 0 no symptom to 10 worst possible symptoms.
  A mixed effect regression model with the anxiety scores from the ESAS will be fit to assess association between groups and outcomes. The study team will also test for time effects and for a group by time interaction effect.
Pre-BMAB Questionnaire | Within fifteen minutes pre-BMAB
  A survey will be offered to those who decline to enroll in order to further understand why they chose not to participate in the study. Survey consists of 6 likert-style questions scored from 0 to 4, with higher scores indicating more agreement with statements. Scores range from 0 to 24, with higher scores indicating more agreement with the statement.
  Also includes an opportunity to list "other reasons" for not participating
Post-BMAB Questionnaire | Within fifteen minutes post-BMAB
  A survey will be offered to those who enroll on the study to fully understand their experience with LOA treatments, assess patients' satisfaction with the lavender oil treatment, if they would be interested in lavender oil for future BMA, and their experience in the clinical trial as a whole. These questions will be based on the Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - General (FACIT-TS-G) questionnaire and tailored to lavender oil aromatherapy.
  Survey consists of 2 sections of 4 likert-style questions (agreement and satisfaction, respectively), with each question scored from 0 to 4 (total section score ranges from 0 to 32, with higher scores indicating more agreement or satisfaction.
  3 additional yes/no/maybe questions relating to whether participant experience and satisfaction follow.
  One additional open-ended question leaves room fore participants to enter other comments.
Percent of patients that decline the study | Within fifteen minutes pre-BMAB
  Feasibility, as measure by percent of patients that decline the study
  If >50% of patients agree to participate and if >50% are able to complete the lavender oil treatment, the study will be determined feasible
Percent of participants completing the study | Within fifteen minutes post-BMAB
  Completion rate, as measured by percent of participants completing the study with 95% confidence intervals, with "completion" defined as receiving lavender oil treatments as described. Each participant will be assigned one of the following categories:
  1. completed treatment course
  2. incomplete treatment course
  9) unknown (not assessable, insufficient data)
  If >50% of patients agree to participate and if >50% are able to complete the lavender oil treatment, the study will be determined feasible
length of time of the BMAB procedure | Within fifteen minutes post-BMAB
  length of time of the BMAB procedure will be compared between LOA versus SOC

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, MD, Principal Investigator — University Hospitals at Cleveland Medical Center